CLINICAL TRIAL: NCT01489124
Title: The Population Pharmacokinetics of Imipenem in Patients With Ventilator-associated Pneumonia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sutep Jaruratanasirikul (Other)
Collaborators: Prince of Songkla University (Other)
Responsible Party: Sponsor-Investigator, Sutep Jaruratanasirikul, Principal Investigator, Prince of Songkla University
Organization: Prince of Songkla University (Other)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: IMI-50-372-028
Record Dates: First submitted 2011-11-23; First posted 2011-12-09 (Estimated); Last update posted 2011-12-09 (Estimated); Status verified 2011-12

CONDITIONS: Ventilator-Associated Pneumonia
Keywords: Infection; Imipenem; Ventilator-Associated Pneumonia; pharmacokinetic; pharmacodynamic
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Infections | interventions — Imipenem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 0.5 g of imipenem by 0.5-hr infusion (Experimental): 0.5 g of imipenem every 6 hrs administrated by 0.5-hr infusion for 3 days
  Interventions: Drug: Imipenem
- 0.5 g of imipenem by 2-hr infusion (Experimental): 0.5 g of imipenem every 6 hrs administrated by 2-hr infusion for 3 days
  Interventions: Drug: Imipenem
- 1 g of imipenem by 2-hr infusion (Experimental): 1 g of imipenem every 6 hrs administrated by 2-hr infusion for 3 days
  Interventions: Drug: Imipenem

INTERVENTIONS:
Drug: Imipenem — 0.5 g of imipenem every 6 hrs administrated by 0.5-hr infusion for 3 days
  Other Names: Imipenem (Tienam)
  Arms: 0.5 g of imipenem by 0.5-hr infusion
Drug: Imipenem — 0.5 g of imipenem every 6 hrs administrated by 2-hr infusion for 3 days
  Other Names: Imipenem (Tienam)
  Arms: 0.5 g of imipenem by 2-hr infusion
Drug: Imipenem — 1 g of imipenem every 6 hrs administrated by 2-hr infusion for 3 days
  Other Names: Imipenem (Tienam)
  Arms: 1 g of imipenem by 2-hr infusion

SUMMARY:
This is prospective, randomized and crossover design to assess the pharmacokinetic and pharmacodynamics of three regimen.

* 0.5-hr infusion of imipenem 0.5 g every 6 hrs
* 2-hr infusion of imipenem 0.5 g every 6 hrs
* 2-hr infusion of imipenem 1 g every 6 hrs

Clinical and laboratory data such as Age,Sex, Body weight, CBC, Electrolyte, Vital signs, APACHE II score, BUN, Cr, Sample and Blood culture will be collected.

Nine patients will be enrolled in this study. After completion of the imipenem therapy for 3 days in this study, all patients will receive other sensitive antibiotics to eradicate their bacterial infections.

Blood samples (approximately 3 ml) will be obtained by direct venepuncture at the following time: 0, 0.5, 1, 2, 3, 4, 5 and 6 after 4th dose of imipenem.

Concentration of imipenem in plasma will be measured by HPLC method. Then, the data will be simulated in Monte Carlo technique (Computer model) to get PK/PD index (40%T>MIC) and reported to % PTA (Probability Target Attainment) and %CFR (Cumulative Faction Response).

DETAILED DESCRIPTION:
Introduction: Ventilator-associated pneumonia (VAP) is a common cause of nosocomial infection with a high mortality rate. In the current era of increasing highly resistant pathogens in nosocomial infections, the empirical treatment of these organisms is becoming more difficult and only a few novel antimicrobial agents are currently in development with activity against these highly resistant Gram negative bacilli infections. Imipenem, a carbapenem antibiotic, is a β-lactam antibacterial agent with a broad spectrum of activity against both Gram positive and Gram negative bacteria. This agent is still one of the most commonly used antibiotics for empirical therapy of highly resistant nosocomial infections in VAP. In common with other β-lactams, imipenem exhibits primarily time dependent killing and increasing the concentration of this agent does not necessarily increase the rate and extent of bacterial killing. Therefore, the time that concentrations in serum are above the MIC (T>MIC) is the pharmacokinetic/pharmacodynamic (PK/PD) index that correlates with efficacy. Pharmacodynamic analysis can be applied to imipenem dosages to increase the likelihood of optimal exposure and achieve good clinical responses in patients with VAP. Previous studies we performed found that a 2 h infusion of carbapenem antibiotics gave greater values for T>MIC than a 0.5 h infusion. Therefore, in an attempt to improve the efficacy of the present β-lactam antimicrobial agents such as imipenem, a prolonged infusion would be the appropriate mode for administration to promote the maximal bactericidal effect.PK changes have been found for several hydrophilic antimicrobial agents in critically ill patients. Drug dispositions are altered in this patient population when compared with healthy subjects leading to fluctuations of plasma concentrations. Therefore, the aim of this study was to assess the PD of imipenem in VAP patients, comparing administration by 0.5 h infusion or 2 h infusion.

Objectives: To assess the pharmacokinetic and pharmacodynamics of three regimen as below.

i) 0.5-hr infusion of imipenem 0.5 g every 6 hrs ii) 2-hr infusion of imipenem 0.5 g every 6 hrs iii) 2-hr infusion of imipenem 1 g every 6 hrs

Drug preparation:Imipenem will be reconstituted with 100 ml saline solution according to the manufacturer's guidelines

Study design: This is prospective, randomized and crossover design to assess

Each patients will receive doripenem in 3 regimens consecutively:

i) 0.5-hr infusion of imipenem 0.5 g every 6 hrs ii) 2-hr infusion of imipenem 0.5 g every 6 hrs iii) 2-hr infusion of imipenem 1 g every 6 hrs

Nine patients will be enrolled in this study. After completion of the imipenem therapy for 3 days in this study, all patients will receive other sensitive antibiotics to eradicate their bacterial infections.

Sample collections: Blood samples (approximately 3 ml) will be obtained by direct venepuncture at the following time: 0, 0.5, 1, 2, 3, 4, 5 and 6 after 4th dose of imipenem. All blood samples will be allowed to clot and then centrifuged at 2,000g. The serum obtained will be stored at-80°C until analysis.

Imipenem assays by HPLC method e performed at Department of Medicine, Faculty of Medicine.

Clinical and laboratory data such as Age,Sex, Body weight, CBC, Electrolyte, Vital signs, APACHE II score, BUN, Cr, Sample and Blood culture will be collected.

Duration of study: Patients will receive imipenem for 3 days

Pharmacokinetic and pharmacodynamic analysis: Concentration of imipenem in plasma will be measured by HPLC method and simulated in Monte Carlo technique (Computer model) to get PK/PD index (40%T>MIC) and reported to % PTA (Probability Target Attainment) and %CFR (Cumulative Faction Response).

Sample Size: Nine patients with VAP will be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years
* Patients are intubated and receiving mechanical ventilation.
* Patients have clinical suspicion of VAP with Gram negative bacilli infections, defined by a new and persistent infiltrate on chest radiography associated with at least one of the following: purulent tracheal secretions, temperature of 38.3°C or higher or a leucocyte count higher than 10000 cells/mm3.
* Expected life expectancy ≥ 3 days

Exclusion Criteria:

* Patients have documented hypersensitivity to imipenem or other carbapenems.
* Patients have an estimated creatinine clearance < 60 ml/min
* Patients are in circulatory shock (defined as a systolic blood pressure of < 90 mmHg).
* Patients are pregnant.
* Pretient receive imipenem for 2 weeks before randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Efficacy of imipenem administration by a 0.5 h and 2 h infusion | At 0, 0.5, 1, 2, 3, 4, 5 and 6 hours after 4th dose of imipenem.
  Concentration of imipenem in plasma will be simulated in Monte Carlo technique (Computer model) to get PK/PD index (40%T>MIC) and reported to % PTA (Probability Target Attainment) and %CFR (Cumulative Fraction Response).

CONTACTS AND LOCATIONS:
Overall Officials: Sutep Jaruratanasirikul, MD, Principal Investigator — Prince of Songkha
Locations (1):
- Prince of Songkla University, Hat Yai, Changwat Songkhla, Thailand